CLINICAL TRIAL: NCT05190276
Title: Incidence and Risk Factors of Symptomatic Epidural Hematoma After Cervical Spine Surgery:a Retrospective Study
Brief Title: Incidence and Risk Factors of Symptomatic Epidural Hematoma After Cervical Spine Surgery
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LM2020298
Record Dates: First submitted 2021-07-01; First posted 2022-01-13 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2021-07

CONDITIONS: Symptomatic Epidural Hematoma After Cervical Spine Surgery
Keywords: epidural hematoma; cervical spine surgery; Risk factors
MeSH Terms: conditions — Hematoma, Epidural, Spinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The hematoma group: with symptomatic epidural hematoma after surgery
- The control group: without symptomatic epidural hematoma after surgery

SUMMARY:
The incidence and correlation of symptomatic epidural hematomas after cervical spine surgery was reviewed and analyzed, then it will provide reference to avoid the occurrence of this complication for the future clinical work.

DETAILED DESCRIPTION:
43 patients with symptomatic epidural hematoma after cervical spine surgery were enrolled in the Peking University Third hospital from January, 2009 to February, 2017. 86 patients without symptomatic epidural hematoma after cervical spine surgery during the same period were randomly selected as the control group. Demographic information (including gender, age, previous history, smoking history, etc.)，disease parameters (diagnosis, mJOA(modified Japanese Orthopaedics association) score, NDI(neck disability index) score)，laboratory and imaging parameters (including platelet, coagulation function, albumin, and OPLL)，segments，treatment parameters (surgical method, number of surgical segments, operative time, intraoperative blood loss, anesthesia time, whether to use implants) and postoperative conditions (including the time of hematoma occurrence, diagnostic method, emergency debridement operation time, patient improvement before and after debridement) were collected.Firstly, risk factors for symptomatic epidural hematoma after cervical surgery were selected by univariate analysis,then independent risk factors were screened by multiple Logistic regression analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinically and radiologically confirmed cervical spondylosis.
* Cervical spine surgery was performed in our hospital

Exclusion Criteria:

* Cervical trauma combined with fracture and dislocation.
* Cervical cancer.
* Cervical spine infection
* Upper cervical spine surgery alone

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent cervical spine surgery in the Department of Orthopedics, Peking University Third Hospital between January 2009 and February 2019
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2019-03-02 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
VAS(visual analogue pain scale) | 3 months after surgery
  visual analogue pain scale, to evaluate patients' pain, form 0 to 10. more scores means more pain
Frankel score | 3 months after surgery
  Postoperative Neurological Function，From A to E. Score A means complete paralyzed and E means no paralyzed
mJOA | 3 months after surgery
  Postoperative Neurological Function, modified Japanese orthopaedics association, From 0 to 17 scores. More scores mean better recovery after surgery. Score 0 means the most severe symptoms.

SECONDARY OUTCOMES:
whether patients occur hematoma after surgery | From post operation immediately till 3 months after surgery
  whether patients occur hematoma after surgery
whether patients need emergency debridement | From post operation immediately till 3 months after surgery
  whether patients need emergency debridement caused by hematoma
the place that occur hematoma | From post operation immediately till 3 months after surgery
  the place that occur hematoma, to locate the place of hematoma from post operation immediately till 3 months after surgery
postoperative neurological recovery after treatment of hematoma | From post operation immediately till 3 months after surgery
  To record neurological recovery after treatment of hematoma from post operation immediately till 3 months after surgery, use modified Japanese Orthopaedics association

IPD SHARING:
Plan to Share IPD: No